CLINICAL TRIAL: NCT04243018
Title: Feasibility Pilot Randomised Control Trial for Brief Acceptance and Commitment Therapy (ACT) Intervention for Adults Experiencing Homelessness to Enhance Well-Being and Mitigate the Deleterious Effects of Shame and Self-Stigma
Brief Title: Feasibility Trial of an Acceptance and Commitment Therapy Intervention for Individuals Experiencing Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HS19-13Murthy-McHugh
Record Dates: First submitted 2019-09-24; First posted 2020-01-27 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-04

CONDITIONS: Shame; Stigma, Social; Well-Being
Keywords: Shame; Self-Stigma; Homelessness; Well-being
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental): Acceptance and Commitment Therapy Intervention to improve well-being and reduce the negative effects of shame and self-stigma in a population of adults experiencing homelessness.This will involve participating in two sessions, lasting two and a half hours each, over a period of two weeks. Well-being will be promoted in each session by targeting core processes of the ACT model including acceptance, cognitive defusion, mindfulness, flexible perspective taking, values clarification and committed action. In addition participants will be provided with an acceptance and commitment training workbook. The workbook will foster core processes of the ACT model through psycho-education, daily exercises, tips and tools.
  Interventions: Behavioral: Acceptance and Commitment Therapy Group Treatment
- Peer Support Group (Active Comparator): This peer support group will involve discussing themes around experiencing homelessness, shame and stigma and will be facilitated by an experienced peer support group leader.This will involve participating in two sessions, lasting two hours each, over a period of two weeks.
  Interventions: Behavioral: Peer Support Group

INTERVENTIONS:
Behavioral: Acceptance and Commitment Therapy Group Treatment — The intervention presents, a mixture of instruction, discussion, and the use of metaphor and experiential activities designed to sensitise participants to the effects of self-stigma and shame on how they live their lives. This training condition provides instruction and experiences that train participants to notice, and then to override, the very human tendency to categorise and then avoid aversive thoughts and feelings and the people and situations that evoke them. The acceptance and commitment training condition will cover the following topics: (a) introduction to enacted and self-stigma (b) cognitive defusion/behavioural flexibility (c) acceptance vs. avoidance and control of emotions and thoughts and (d) values and committed action.
  Arms: Acceptance and Commitment Therapy
Behavioral: Peer Support Group — The peer support group will allow participants to share and discuss experiences related to their experiences of homelessness, shame and stigma. The group will be facilitated by an expert in facilitating peer support groups with marginalised populations.
  Arms: Peer Support Group

SUMMARY:
The current project's overall aim is to develop and evaluate the feasibility and preliminary efficacy of an ACT intervention to promote psychological well-being and mitigate the deleterious effects of shame and self-stigma in people experiencing homelessness. This project will advance current knowledge using systematic and empirical methodology to develop and evaluate the benefits of a group-based ACT intervention, which to date has not been explored with this population.

DETAILED DESCRIPTION:
On average homeless persons have higher rates of childhood and adult adversity, challenging behaviour, substance and alcohol misuse, poor educational, occupational achievement, co-morbid physical and mental illness. In mental health, services delivered on the basis of address can struggle to mount a satisfactory response to the needs of homeless persons. Many homeless persons rely on emergency department visits or inpatient hospitalizations for health care. When admitted to hospital, they have longer stays with higher costs. With the rates of homelessness increasing in both national and international contexts coupled with the several barriers to accessing mainstream health services, the development of brief, cost-effective interventions, that address comorbidity of various mental illnesses and substance abuse is necessary.

In addition, individuals who have experienced homelessness can have their growth and development curtailed by applying a punitive, shame based, and defeatist perspectives to their own goals and values in life. Direct acts or discrimination, as well as diminished opportunities offered to people experiencing homelessness, can be understood as a manifestation of public stigma. Labelling someone as "homeless" or an "addict" tends to activate common stereotypes such as thinking that the person is likely to be unreliable, deceitful, or weak, among other stereotypes. This often leads to some sort of social sanction or devaluation, reducing the probability of the person being hired, or being trusted as a parent, friend, or lover.

People who identify with a stigmatised group often internalise the stereotypes associated with that group. In addition, the effects of enacted stigma, the emotional and cognitive barriers erected by the individual experiencing homelessness in response to perceived or experienced stigma, can also serve to obstruct access to opportunities. The person may self-identify as a loser, being damaged goods, or always hurting others. Attachment to these self-conceptions entails giving up on important and valued life directions. These are manifestations of self-stigma. Studies of individuals with serious mental illness and co-occurring disorders have shown that self-stigma is associated with delays in treatment seeking or avoidance of treatment, diminished self-esteem/self-efficacy, increased mental health symptoms, and lower quality of life. Therefore, it is imperative that interventions actively address and aim to mitigate the deleterious effects of shame and self-stigma.

Assertive Community Treatment and case-management interventions have been proven moderately effective in improving mental and physical health outcomes for homeless populations, however, the resources and expertise required to run such interventions are; unavailable to most sectors and communities, time consuming and normally used on an individual case basis, leaving large portions of this population untreated. Research into brief psychological interventions with the homeless population has revealed promising effects, however, these interventions often target specific sub-populations, chose to focus on one aspect of recovery such as substance abuse and do not address comorbidity of illness.

The Acceptance and Commitment Therapy(ACT) model is compatible with conceptualisations of recovery from severe mental illness (defined as "living a satisfying, hopeful and contributing life even with limitations caused by the illness"; and "having a sense of purpose and direction"). From an ACT perspective 'addictive-', 'depressive-', 'anxiety'- and "stress-' behaviours might share the same function; and those with high levels of comorbidity, such as the homeless population might therefore be treated using an ACT.

The focus on specific cognitive behavioural processes of mindfulness, acceptance, distancing, and values-based action makes ACT interventions typically brief and have been proven to be effective after a single session and mediation studies suggest that the positive clinical effects of ACT are achieved by changing these targeted psychological processes.

A two-arm feasibility pilot randomised control trial will be conducted to investigate differences in the proposed outcome variables between participants assigned to a group-based ACT intervention and those assigned to peer support group. A process level investigation will also be used to investigate the feasibility of conducting a full scale RCT with the population.

ELIGIBILITY:
Inclusion Criteria:

- Service Users: Individuals who are currently experiencing or have experienced homelessness in the past year.

Over 18 and under 65.

- Service Providers: Have been working with homeless services for over a year, in close contact with service users. Over 18 and under 65.

Exclusion Criteria:

* Participants with severe mental health issues- Currently experiencing suicidal ideation or active psychosis
* Participants with serious cognitive impairments
* Participants with below conversational level proficiency in English

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Internalised Shame Scale (Cook, 1996) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  30-item measure that assess shame proneness and internalised shame. It also contains a 6-item self-esteem scale.Respondents must rate each self-statement on a Likert-type scale from 0 to 4, with each number anchored to the words, "Never", "Seldom", "Sometimes", "Often", and "Almost Always", respectively. Higher scores indicate more problematic levels of internalised shame. Higher scores on the self-esteem sub-scale indicate positive self-esteem. Scores of the sub-scales are summed to provide a total score for internalised shame.
Self-Stigma Scale- Short (Mak & Cheung, 2010) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  a 9-item measure that is conceptualised along three psychological dimensions (viz., self-stigmatising cognition, affect, and behaviour), and corresponds to cognitive-behaviour theory.Each item asks the respondents to rate their agreement on a 4-point Likert scale from 1 (strongly disagree) to 4 (strongly agree). Higher score on the SSS-S represents a higher level of self-stigma.
World Health Organisation- Five Well-Being Index (WHO, 1998) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  5-item short self-reported measure of current mental well-being.
CompACT Scale (Francis, Dawson, & Moghaddam, 2016) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  23-item measure assessing Acceptance and Commitment Therapy specific outcomes, psychological flexibility, valued action, openness to experience, and behavioural awareness.
Identifying Levels of Treatment Engagement | 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  Semi-structured interviews will also be conducted with a service user from each group and with service providers, this done in order to assess treatment engagement and also inform a process level investigation.
Therapist Fidelity and Adherence | 3-months post-baseline (follow-up)
  Treatment fidelity will be assessed post-intervention by 2 independent reviewers (members of the Contextual Behavioural Sciences lab in UCD). This will involve reviewers listening to the same 10-minute recording from each session and listing the ACT processes they can identify within the 10-minute recording. With the aim of achieving a minimum of 70% consensus between reviewers. Therapists will also have to write down what exercises were used to teach each of the ACT processes post-intervention for each session and will be assessed by the independent reviewers to assess protocol adherence; were all of the ACT processes taught and were the exercises in the protocol used.
Study Feasibility Interviews | 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  Service users will be asked about the practicalities of participating the study (e.g. experience of answering questionnaires), experiences of the group, how the intervention has impacted the environment in the shelter, what they found most beneficial, recommendations for improvements, and engagement with intervention and the use of skills learned.Service provider interviews will explore, feasibility of the intervention, resource management, staff-researcher communication and the intervention. Results from these interviews, therapist adherence and fidelity, and analysis of retention and attrition will be the process-based outcomes from the study.
Participant Retention and Attrition | Post-completion of data collection an average of one-year
  Percentage of participants retained at 8-week follow-up. Percentage of participants who attended each session and data collection point
Client Satisfaction Questionnaire-8 (CSQ-8; Attkisson, Hargreaves & Nguyen, 1978) | 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  8-item self-report statement of satisfaction with health and human services.

SECONDARY OUTCOMES:
Cognitive Fusion Questionnaire (Gillanders et al., 2014) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  seven items rated on a 7-point scale of 1 (never true) to 7 (always true) designed to measure the relationship a person has with his or her own thoughts and beliefs
Hospital Anxiety and Depression Scale (HADS; Zigmond, & Snaith 1983) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  A self-report rating scale of 14 items, designed to measure anxiety (HADS-A) and depression (HADS-D), with each subscale consisting of 7 items. It consists of two sub-scales yielding a separate score for anxiety and depression.
Present Moment Awareness Subscale of the Philadelphia Mindfulness Scale (Cardaciotto, Herbert, Forman, Moitra & Farrow, 2008) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  10-item self-report questionnaire that measures a key constituent of mindfulness
Self-Compassion Scale-Short Form (Raes, pommier, Neff, & Van Gutcht, 2011) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  12-item measure that examines the relation of self-compassion to positive psychological health and the five-factor model of personality.
Valuing Questionnaire (Smout, Burns & Christie, 2014) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  10-item measure that assesses the degree of personal values enactment "during the past week." Items are rated on a 7-point scale ranging from 0 (not at all true) to 6 (completely true).
Mental Health Continuum - Short Form (Keyes, 2005) | Baseline; 1-month post-baseline (post-intervention); 3-months post-baseline (follow-up)
  14-item measure of positive mental health consisting of three sub-scales: Emotional well-being, psychological well-being, and social well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Louise McHugh, PhD, Principal Investigator — University College Dublin
Locations (3):
- Ireland (3):
  - Merchants Quay Ireland, Dublin
  - Focus Ireland, Dublin
  - Peter McVerry Trust, Dublin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will become available post publication of the study. This data will be available indefinitely.